CLINICAL TRIAL: NCT02162953
Title: Development of Induced Pluripotent Stem Cells From Patients With Best Disease and Other Inherited Retinal Degenerative Diseases.
Brief Title: Stem Cell Models of Best Disease and Other Retinal Degenerative Diseases.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Alan D. Marmorstein, Ph.D., Professor of Ophthalmology,, Mayo Clinic
Other Study IDs: 13-008089; U01EY030547 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Retinal Disease; Bestrophinopathy; Best Vitelliform Macular Dystrophy; Adult Onset Vitelliform Macular Dystrophy; Autosomal Dominant Vitreoretinalchoroidopathy
Keywords: eye disease; retinal; best1
MeSH Terms: conditions — Retinal Diseases; Bestrophinopathy; Vitelliform Macular Dystrophy; Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (10 ml) for DNA/RNA extraction
  Dermal Tissue from Skin punch biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Autosomal recessive bestrophinopathy (ARB) is one of 5 blinding eye diseases caused by mutations in the gene BEST1. These diseases, collectively termed "bestrophinopathies" include ARB, Best vitelliform macular dystrophy (BVMD), adult-onset vitelliform dystrophy (AVMD), autosomal dominant vitreoretinalchoroidopathy (ADVIRC) and retinitis pigmentosa (RP) .

Objective: To collect DNA/RNA and skin samples from individuals with ARB or other diseases due to mutations in the gene BEST1. These models will be used to identify and test therapeutic approaches to treating these diseases.

Design: Study involves a one time donation of a skin punch biopsy and whole blood. Once the skin biopsy is obtained, skin fibroblasts will be isolated, which will be reprogrammed into iPSCs. RPE cells will be derived from the iPSCs

DETAILED DESCRIPTION:
The PI on this proposal has been studying BEST1 and the protein encoded (Best1) since its discovery in 1998. Best1 is an integral membrane protein that in the eye is expressed only by retinal pigment epithelial (RPE) cells where it is localized to the basolateral plasma membrane.

Methods: Once a subject has been identified as a potential candidate, a study coordinator will meet with the subject, to discuss the study prior to sample collection. The study coordinator will review the consent form with the subject and spend as much time as necessary answering any questions. Once the subject has signed the consent form, study procedures will begin.

Following the consent process, a skin sample will be obtained from subjects using a (4mm) dermal punch biopsy method. This will be accomplished in a single visit to the Regenerative Medicine Consult Service or other approved clinical examination room. A suture may need to be placed following this skin biopsy. A health care provider (either at Mayo Clinic or a local health care provider's office) can remove the stitches, or the subject can remove them with a provided disposable suture removal kit.

Subjects will also be asked to undergo venipuncture; all subjects will be asked to have the venipuncture and have the option to refuse. 10ml of blood will be collected for RNA and DNA extraction.

Once the skin biopsy is obtained,skin fibroblasts will be isolated, which will be reprogrammed into iPSCs. RPE cells will be derived from the iPSCs.

Remuneration: If subjects make a special trip only for the research procedures, they may be reimbursed for travel expenses including: airfare, mileage, parking, and hotel. In order to receive reimbursement, they must provide a copy of the original receipts for those expenses. Reimbursement will not exceed $1000.00.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been diagnosed on the basis of genotyping with a bestrophinopathy.
* Patient must be willing to provide a skin biopsy from which we will generate iPSCs.
* For pediatric patients, parents must be willing to donate skin biopsies as well.

Exclusion Criteria:

* Children under the age of 5
* Patients exhibiting secondary ophthalmic disorders that are not typically associated with the bestrophinopathies may be excluded.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children (as well as their parents) and adults with mutations in the gene BEST1 resulting in one of the five bestrophinopathies.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of iPS cells successfully differentiated into RPE cells | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alan D. Marmorstein, Ph.D., Principal Investigator — Mayo Clinic; Raymond Iezzi, M.D., Principal Investigator — Mayo Clinic; Sophie J. Bakri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
All samples will be de-identified and given a code while stored and used in research. IPD available to other researchers might include age, gender, genetic mutation and diagnosis. No other information will be shared.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials